CLINICAL TRIAL: NCT06167291
Title: Phase II Randomized-registry Embedded Study of Lymphoscintigraphy for Oropharyngeal Neoplasms to Enable Risk-adapted Nodal Guidance for Robotic Surgery and/or Radiotherapy (LONE-RANGR2)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0915; NCI-2023-10400 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Oropharyngeal Neoplasms; Robotic Surgery and/or Radiotherapy; Lymphoscintigraphy
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1- Ipsilateral (Experimental): Participants with ipsilateral-only drainage (Arm 1- Ipsilateral) will be randomized to assign definitive ipsilateral RT (without concurrent chemotherapy) -vs- ipsilateral surgery (TORS/ND).
  Interventions: Radiation: Arm 1- Ipsilateral

INTERVENTIONS:
Radiation: Arm 1- Ipsilateral — Given by I-RT

SUMMARY:
To test a new radiation treatment design based on where your cancer is located. Most participants with oropharyngeal cancer are treated with radiation to both sides of the neck. However, for participants with oropharyngeal cancer on one side of the neck, receiving radiation to both sides of the neck may result in increased side effects and radiation exposure. This study is testing the safety and effectiveness of an approach that involves radiation to only one side of the neck in an effort to reduce the overall amount of radiation given and decrease the amount of side effects you may experience.

DETAILED DESCRIPTION:
Primary Objectives

To determine whether:

1. Omission of the contralateral neck cancer treatment is safe and toxicity-sparing for participants with well lateralized oropharyngeal HNSCC undergoing definitive or PORT radiation. This will be demonstrated by acceptably low contralateral neck failures (<15%)

Secondary Objectives

To determine:

1. the relative difference in symptom burden, as measured by the MDASI_HN area-under-the-toxicity curve (AUC), for initial surgical and initial non-surgical therapy cohorts.
2. Whether omission of the contralateral neck in radiotherapy planning as definitive of PORT treatment for well-lateralized oropharyngeal tumors will impact symptom burden as measured by MDASI AUC, Grade 2 or higher CTCAE v5.0 toxicity, swallow function, and/or feeding tube rates and dependency.
3. Risk adapted therapy approaches lead to differences in distant-metastasis-free survival (DMFS), ipsilateral neck failure, primary site failure, and whether salvage therapy for contralateral neck failures is feasible and effective compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histopathologically-proven p16+ and/or HPV+ HNSCC of the base of tongue or faucial tonsil
* cT1-2N0-1 per AJCC 8th edition staging.
* Tumor does not cross midline, and must be >1cm from midline
* For tonsil tumors, the primary may extend onto the palate or into the BOT but still be >1cm from midline
* No evidence of contralateral neck disease on contrast MRI, CT Head/Neck, PET/CT, or lymphoscintigraphy nor retropharyngeal lymphadenopathy.
* Able to undergo lymphoscintigraphy procedure
* No contraindications for SLNM, adjuvant chemotherapy, RT nor adjuvant/definitive radiotherapy.
* ECOG 0-1
* Age >18 years
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Previous HN Cancer except small skin cancers.
* Any retropharyngeal lymphadenopathy on either MRI, CT, or PET/CT
* Contralateral neck nodal disease radiographically detected per routine diagnostic imaging or SPECT-CT.
* Distant metastatic spread at the time of inclusion
* Chemotherapy or surgery (for the present tumor), prior to inclusion.
* Previous radiation treatment in the head and neck region, for any reason, except for cutaneous lesions that would not lead to overlap with definitive bilateral neck irradiation
* Recurrent or second primary tumor in the head and neck region
* Non-tongue base or non-faucial tonsil primaries
* Prior history of regionally advanced or distant spread cancers
* Pregnancy or no active contraception for pre-menopausal women
* Known hypersensitivity to iodine or nanocolloid injection
* Having any condition (physical, mental, sociological) that interferes with the informed consent procedure and follow-up schedules Has a diagnosis of active scleroderma, lupus, or other rheumatologic disease which in the opinion of the treating radiation oncologist precludes safe radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2027-12-09 (Estimated); Study Completion 2027-12-09 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: David Rosenthal, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org